CLINICAL TRIAL: NCT02385305
Title: The Effect of Pressure Support Ventilation on Minute Alveolar Ventilation and End-tidal Carbon Dioxide in Anesthetized Spontaneously Breathing Subjects
Brief Title: The Effect of Pressure Support Ventilation on Spontaneous Breathing in Anesthetized Subjects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, MD, PhD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2014P001841
Record Dates: First submitted 2014-12-01; First posted 2015-03-11 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia
Keywords: Pressure support ventilation; respiratory drive; Physiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pressure support ventilation (Other): Usual anesthesia management
  Interventions: Device: Pressure support ventilation by anesthesia machine (Apollo, Dräger)

INTERVENTIONS:
Device: Pressure support ventilation by anesthesia machine (Apollo, Dräger) — Pressure support ventilation will be applied by anesthesia machine (Apollo, Dräger) with pressure support (PS) of 3, 8, 13 and 18 cmH2O in this order, with slope of 1.0 second and no PEEP. The fraction of inspired oxygen will be titrated to achieve SpO2 over 98%. Five minutes will be allowed to achieve equilibrium at each PS level after which an additional recording of one minute of data will be obtained. Once the Pressure support ventilation is completed at 18 cmH2O, ventilation will be carried out in reverse order of PS; 13, 8 and 3 cmH2O of PS.

SUMMARY:
The aim of this prospective study is to determine the effect of pressure support ventilation (PSV) on minute alveolar ventilation (MAV) and end-tidal carbon dioxide (ETCO2) in anesthetized spontaneously breathing subjects by observing alterations of respiratory rate (RR), expiratory tidal volume, MAV and ETCO2 at variable levels of pressure support.

DETAILED DESCRIPTION:
Anesthesia induction will be performed with usual anesthetics without any opioids and followed by the placement of a laryngeal mask airway. Optimal anesthesia level will be maintained with inhalation anesthesia so as to obtain a bispectral index of 30 to 50. Subjects will be ventilated with controlled mechanical ventilation (CMV) by the anesthesia ventilator until the presence of spontaneous breathing can be affirmed. A carbon dioxide/flow sensor (Adult Combined CO2/Flow Sensor; Novametrix medical systems INC., Wallingford, CT) will be placed between the LMA and the breathing circuit. The sensor will be connected to a noninvasive cardiac output monitor (NICO; Noninvasive Cardiopulmonary management System, model 7300; Respironics Corp., Murrysville, PA). NICO data (end-tidal CO2 (ETCO2), tidal volume and flow waveforms) will be recorded and stored on a personnel computer. At the start of surgery, the anesthesia care provider will administer opioids to control nociceptive stimuli from surgery. Figure 2 shows the procedural course of the study. Once spontaneous breathing is observed, PSV will be applied with pressure support (PS) of 3, 8, 13 and 18 cmH2O in this order, with slope of 1.0 second and no PEEP. The fraction of inspired oxygen will be titrated to achieve SpO2 over 98%. Five minutes will be allowed to achieve equilibrium at each PS level after which an additional recording of one minute of data will be obtained. Once the PSV is completed at 18 cmH2O, ventilation will be carried out in reverse order of PS; 13, 8 and 3 cmH2O of PS. If at any point in the course of the study the subjects ETCO2 is higher than 60 mmHg, obvious body motion is observed or abnormal vital signs [NIBP; >160/90 mmHg or <80/50 mmHg, HR; >100 mmHg or <40 mmHg, SpO2; <94% at a given fraction of inspired O2] occur, the study will be terminated and routine care will be provided.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status classification I or II
2. Expected to be ventilated with a laryngeal mask airway (LMA)
3. Expected to have anesthesia titrated to insure continued spontaneous breathing

Exclusion Criteria:

1. Patients whose surgery will last less than 70 minutes
2. Obese patients with BMI 30 kg/m2 or higher
3. Patients who will have thoracic or abdominal surgery
4. Patients with gastro-esophageal reflux disease
5. Patients who will needed muscle relaxants or are expected to require controlled ventilation during surgery
6. Patients with chronic obstructive pulmonary disease or asthma
7. Patients with neuromuscular disease or presenting with increased intracranial pressure
8. Patients with major cardiovascular disease, or cerebral vascular disease
9. Abnormal vital signs on the day of admission for surgery [heart rate (HR); >100 bpm or <40 bpm, Noninvasive blood pressure (NIBP); >180/100 mmHg or <90/60 mmHg or transcutaneous oxyhemoglobin saturation (SpO2); <94%] that are not correctable with his or her routine medication or commonly used pre-operative medication
10. Pregnant women and women less than one month post-partum. Pregnancy will be ruled out by careful history and physical examination. If history is equivocal, the subject will be excluded unless a negative pregnancy test is obtained
11. Emergent cases
12. Chronic opioid use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
End-tidal carbon dioxide measured by Capnograph monitor | 0, 5, 10, 15, 20, 25, 30 and 35 min after the initiation of PSV
  end-tidal carbon dioxide (mmHg): this assessment relies on multiple measurements over time and the Time Frame includes multiple time points

SECONDARY OUTCOMES:
Respiratory rate measured by Respiratory monitor | 0, 5, 10, 15, 20, 25, 30 and 35 min after the initiation of PSV
  respiratory rate (breath/min): this assessment relies on multiple measurements over time and the Time Frame includes multiple time points
Expiratory tidal volume measured by Respiratory monitor | 0, 5, 10, 15, 20, 25, 30 and 35 min after the initiation of PSV
  expiratory tidal volume (ml): this assessment relies on multiple measurements over time and the Time Frame includes multiple time points

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jian, MD, PhD, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Background] Pattinson KT. Opioids and the control of respiration. Br J Anaesth. 2008 Jun;100(6):747-58. doi: 10.1093/bja/aen094. Epub 2008 May 1. PMID 18456641
- [Background] Yamanaka T, Sadikot RT. Opioid effect on lungs. Respirology. 2013 Feb;18(2):255-62. doi: 10.1111/j.1440-1843.2012.02307.x. PMID 23066838